CLINICAL TRIAL: NCT04848077
Title: STEPWISE Parkinson: A Smartphone Based, Titrated Exercise Solution for Patients With Parkinson's Disease in Daily Life
Brief Title: STEPWISE Parkinson: A Smartphone Based Exercise Solution for Patients With Parkinson's Disease
Acronym: STEPWISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Massachusetts General Hospital (Other); Hogeschool van Arnhem en Nijmegen (HAN) (Unknown); Canisius-Wilhelmina Hospital (Other); IJsfontein Health BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL75501.091.20
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-11

CONDITIONS: Movement Disorders; Parkinson Disease
Keywords: Physical activity; Walking; Exercise; Parkinson Disease; Locomotion; Motivational application
MeSH Terms: conditions — Movement Disorders; Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Very high dose (Experimental): Very large proportional increase in stepcount relative to baseline stepcount.
  Interventions: Behavioral: Step count increase with the use of a motivational smartphone application
- High dose (Experimental): Large proportional increase in stepcount relative to baseline stepcount.
  Interventions: Behavioral: Step count increase with the use of a motivational smartphone application
- Intermediate dose (Experimental): Medium proportional increase in stepcount relative to baseline stepcount.
  Interventions: Behavioral: Step count increase with the use of a motivational smartphone application
- Active controls (Active Comparator): Small proportional increase in stepcount relative to baseline stepcount.
  Interventions: Behavioral: Step count increase with the use of a motivational smartphone application

INTERVENTIONS:
Behavioral: Step count increase with the use of a motivational smartphone application — All participants will be given access to an application installed on the participants' own smartphone: the STEPWISE app. The STEPWISE app will encourage participants to increase their long-term physical activity (1 year). Different treatment arms will receive different physical activity goals. Participants will get feedback and support via the smartphone app, that stimulates them to reach their individual physical activity goal (i.e. target percentage increase in stepcount).

SUMMARY:
The aim of this study is to investigate whether a smartphone app can increase physical activity in patients with Parkinson's Disease in daily life for a long period of time (12 months).

DETAILED DESCRIPTION:
Rationale: Exercise affords health benefits for people with Parkinson's disease (PD), but implementing exercise in daily life remains challenging. Moreover, many training programs are not very scalable. The investigators take an important step forward by developing and studying an innovative and fully decentralized smartphone-based program to increase long-term physical activity in people with PD in daily life.

Objective: The aim of this study is to investigate whether a smartphone app can increase physical activity in PD patients for a long period of time (12 months). The secondary aim is to test the potential group effect on physical fitness, motor- and non-motor symptoms. Thirdly, we aim to investigate whether there is a dose-response relationship between amount of physical activity and physical fitness, motor- and non-motor functioning.

Study design: Double-blind randomized controlled trial.

Study population: A total of 452 Dutch patients with PD who have no other medical conditions that markedly hamper mobility other than PD, no cognitive impairments that make it difficult to use a game on the smartphone and possess a suitable smartphone, will be recruited.

Intervention: Participants will be randomized to a group that will be motivated to increase their physical activity level to a small, medium, large or very large degree with respect to their own baseline level.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD
* Hoehn and Yahr 1-3
* able to understand the Dutch language
* able to walk independently
* equal to or less than 120 minutes of sports/outdoor activities per day (question 5-28 LASA Physical Activity Questionnaire (LAPAQ))
* less than 7,000 steps/day during 1-month baseline (week -4 until 0)

Exclusion Criteria:

* weekly falls in the previous 3 months
* medical conditions that hamper mobility other than PD
* living in a nursing home
* cognitive impairments that hamper use of the motivational app (subjective evaluation by the assessor)
* not in the possession of a suitable smartphone (Iphone 5S or newer with iOS 10 or higher or Android 4.1 or newer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mean change in step count per day | Week -4 until 0 and week 49 until 52
  Mean change in step count per day as measured continuously with the participant's smartphone from baseline (week -4 to 0) to follow-up (week 49-52). Higher scores indicate more physical activity (steps).

SECONDARY OUTCOMES:
Change in physical fitness (6MWT) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline in meters walked during the six minute walk test (6MWT) at week 53 (follow-up). Higher scores indicate better function.
Change in motor- and non-motor aspects of daily living | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline in the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) parts Ib and II at 53 weeks (follow-up). Range 0-80. Higher scores indicate worse function.
Change in physical fitness (VO2max) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline in VO2max in ml/kg/min assessed by a maximal aerobic exercise test on a cycle ergometer at follow-up (week 53). Higher scores indicate better function. Performed in a subgroup of 100 participants.
Change in Parkinson's Disease symptoms (MDS-UPDRS) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline in the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) at 53 weeks (follow-up). Range 0-199. Higher scores indicate worse function.
  Total scores for Parts I, II, III, and IV will also be calculated.
Change in ambulatory capacity (MDS-UPDRS) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline in the sum of 5 MDS-UPDRS questions: walking and balance [question 2.12], freezing [q. 2.13], gait [q. 3.10], freezing of gait [q. 3.11], and postural stability [q. 3.12]). Higher scores imply worse symptoms.
Change in mobility (TUG) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline in the time (seconds) needed to complete the Timed Up and Go Test (TUG) at 53 weeks (follow-up). Higher scores indicate worse function.
Change in balance (Mini-BestTest) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Mini-BestTest at 53 weeks (follow-up).Range 0-28. Higher scores indicate better function.
Change in gait speed (10MWT) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline in gait speed (m/s) as assessed by the 10 meter walk test (10MWT). Higher scores indicate better function.
Change in fear of falling (FES-I) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Dutch version of the Falls Efficacy Scale International at 53 weeks (follow-up). Range 16-64. Higher scores indicate higher fear of falling.
Number of falls and near-falls (monthly fall diary) | Every four weeks after start of the intervention (at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 weeks).
  Number of falls and near-falls reported monthly by the participants in a fall diary drafted according to the European Physiotherapy guideline for Parkinson's Disease.
Change in handgrip strength | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline in hand grip strength (kg) as assessed with a dynamometer (best out of three attempts).
Change in self-reported physical activity level (LAPAQ) | Week -4 (screening), week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Longitudinal Aging Study Amsterdam (LASA) physical Activity Questionnaire (LAPAQ). Higher scores indicate a higher physical activity level.
Change in cognition (MOCA) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Montreal Cognitive Assessement (MOCA) score at 53 weeks (follow-up). Range 0-30. Higher scores indicate better cognition.
Change in depression and anxiety (HADS) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Hospital Anxiety and Depression Scale (HADS) at 53 weeks (follow-up). Range 0-42. Higher scores indicate worse function.
Change in apathy (AES-12PD) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Apathy Evaluation Scale (AES-12PD) at 53 weeks (follow-up). Range 12-48. Higher scores indicate better function.
Change in fatigue (FSS) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Fatigue Severity Scale (FSS) at 53 weeks (follow-up). Range 1-7. Higher scores indicate worse function.
Change in severity of sleep problems and daytime sleepiness (SCOPA-SLEEP) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Scales for Outcomes in Parkinson's Disease - Sleep (SCOPA-Sleep) questionnaire at 53 weeks (follow-up).
Change in autonomic dysfunction (SCOPA-AUT) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Scales for Outcomes in Parkinson's Disease - autonomic questionnaire (SCOPA-AUT) at 53 weeks (follow-up).
Change in Health related quality of life (PDQ-39) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the Health related quality of life (PDQ-39) questionnaire at 53 weeks (follow-up). Range 0-100. Higher scores indicate better function.
Perceived effect of intervention (GPE) | At week 53 (follow-up)
  Perceived effect of intervention as assessed by the Global Perceived effect (GPE) questionnaire (7-point scale) at 53 weeks (follow-up). Range 1-7. Higher scores indicate higher perceived effect.
System Usability (SUS) | At week 53 (follow-up)
  Usability of the STEPWISE application as assessed by the Dutch version of the System Usability Scale (SUS) at 53 weeks (follow-up). Range 0-100. Higher scores indicate better usability.
Perceived physical ability (LIVAS) | Week 0 (baseline) and week 53 (follow-up)
  Change from baseline on the percieved physical ability scale (Lichamelijke Vaardigheden Schaal; LIVAS) at 53 weeks (follow-up). Range 10-50. Higher scores indicate higher perceived phisical ability.

OTHER OUTCOMES:
STEPWISE Parkinson smartphone application data | From baseline (week 0) to follow-up (week 53)
  User data from the STEPWISE smartphone application will be collected, including number of interactions with the app and the total time the application was used.
Adherence to the intervention | From baseline (week 0) to follow-up (week 53)
  Adherence to the study intervention as indicated by the number of days the STEPWISE app was used.
Barriers and motivators to engage in exercise/physical activity at baseline and follow-up | Week 0 (baseline) and week 53 (follow-up)
  Barriers and motivators to engage in exercise/physical activity reported on the self-developed Barriers and Motivators questionnaire at week 0 (baseline) and week 53 (follow-up).
Exploratory measurement of physical acitivity with wearable sensor | From week 0 (baseline) to week 1 and from week 52 to week 53 (follow-up)
  Movement data captured with a 6-axis inertial movement sensor (Axivity AX6).
Parkinson's disease symptoms monitored with the mPower app | Every three months from week 0 (baseline) to week 53 (follow-up)
  Parkinson's disease symptoms monitored remotely with the mPower smartphone app.
Blood-based biomarkers | Week 0 (baseline) and week 53 (follow-up)
  Change in blood-based biomarkers. Assays will be determined before unblinding. Collected for a subgroup of participants (maximum n=135).

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan Bloem, Prof. Dr., Principal Investigator — Radboudumc Department of Neurology
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will make relevant and anonymised data available in a validated database.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the main results of our trial.
Access Criteria: Access to the data is restricted, meaning that researchers who are interested in re-use of the data are asked to contact the central contact person for permission. Approval is given after a signed agreement.

REFERENCES:
- [Derived] Schootemeijer S, de Vries NM, Macklin EA, Roes KCB, Joosten H, Omberg L, Ascherio A, Schwarzschild MA, Bloem BR. The STEPWISE study: study protocol for a smartphone-based exercise solution for people with Parkinson's Disease (randomized controlled trial). BMC Neurol. 2023 Sep 12;23(1):323. doi: 10.1186/s12883-023-03355-8. PMID 37700241

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT04848077/SAP_000.pdf